CLINICAL TRIAL: NCT02607436
Title: Effect of Sarpogrelate, a Serotonin Receptor Antagonist, on Progression of Coronary Artery Disease
Brief Title: Effect of Sarpogrelate, a Serotonin Receptor Antagonist, on Coronary Artery Disease
Acronym: SAGE-CAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1111/139-007
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — sarpogrelate; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sarpogrelate + Aspirin (Experimental): Sarpogrelate as an active drug
  Interventions: Drug: Sarpogrelate; Drug: Aspirin
- Aspirin alone (Active Comparator): Aspirin as an active comparator
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Sarpogrelate — Sarpogrelate
  Other Names: Anplag
  Arms: Sarpogrelate + Aspirin
Drug: Aspirin — Aspirin
  Other Names: Aspirin protect or Astrix

SUMMARY:
This is a prospective interventional study to assess the effect of sarpogrelate compared with aspirin in Korean type 2 diabetic patients with atherosclerosis.

DETAILED DESCRIPTION:
Type 2 diabetes has been increased exponentially, arousing serious economic, social and health repercussions. Also, macrovascular complications of diabetes such as myocardial infarct or stroke have been increased. Individuals with diabetes have a greater risk of cardiovascular disease (CVD), approximately two to four times than that of those without diabetes. Currently, the U.S. Food and Drug Administration requires demonstration that new anti-hyperglycemic agents do not increase cardiovascular risk. The comprehensive and multifactorial management in type 2 diabetes, which includes control of hypertension, dyslipidemia and obesity, is known to significantly reduce the risk of CVD as shown in Steno-2 study. However, most anti-diabetic agents currently used in clinical practice do not seem to provide enough cardiovascular protection.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c ≥ 6.5% at screening visit
* Male or female between 30 and 80 years of age
* Coronary artery stenosis: 10-75% without no evidence of acute coronary syndrome
* No history of previous myocardial infarction

Exclusion Criteria:

* Systolic blood pressure / diastolic blood pressure > 160/110 mmHg
* Congestive heart failure
* Allergy to radiocontrast dye
* Allergy to aspirin or sarpogrelate
* Acute bleeding
* History of ulcer bleeding
* GOT/GPT > 100/100
* Other antiplatelet medication

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease assessed by cardiac computed tomography angiography | 6 months

SECONDARY OUTCOMES:
Coronary artery calcium score assessed by cardiac computed tomography angiography | 6 months
Coronary artery stenosis assessed by cardiac computed tomography angiography | 6 months
Changes of plaque size assessed by cardiac computed tomography angiography | 6 months
Changes of plaque composition assessed by cardiac computed tomography angiography | 6 months
Changes of Ankle-branchial index | 6 months
Changes of pulse wave velocity | 6 months
Glucose metabolism assessed by glycated hemoglobin | 6 months
Lipid metabolism assessed by triglyceride and high density lipoprotein-cholesterol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No